CLINICAL TRIAL: NCT04834284
Title: Decreasing Prehospital Delay to Mechanical Thrombectomy Using a Helicopter Emergency Medical Services Unit
Brief Title: HEMS for Mechanical Thrombectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Sanna Hoppu, MD, PhD, Head of Emergency Medical Services, Tampere University Hospital
Other Study IDs: R20082
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Helicopter Emergency Medical Services (HEMS): Patients transported to the comprehensive stroke centre at least in some part by a HEMS unit
- Ground Emergency Medical Services (GEMS): Patients transported to the comprehensive stroke centre solely by an ambulance

SUMMARY:
Elapsed time from the onset of stroke symptoms to the point of revascularization is the key determinant of the optimal outcome of acute ischemic stroke. Pharmacological treatment is less effective if the thrombus occluding the artery is big enough and mechanical thrombectomy is required to gain recanalization. Mechanical thrombectomy can be done only in comprehensive stroke centres. There are 5 comprehensive stroke centres in Finland which causes regional inequality when it comes to reaching mechanical thrombectomy in a reasonable time limit.

The aims of the study is to measure the effect of dispatching a helicopter emergency medical services unit on the treatment delays of a stroke patient with large vessel occlusion. The HEMS unit is dispatched to both: getting patient directly to the comprehensive stroke centre as well as to interfacility tranfers.

ELIGIBILITY:
Inclusion Criteria:

- all adult patients transferred for mechanical thrombectomy from the South Ostrobothnia Hospital District to the Tampere University Hospital

Exclusion Criteria:

* The neurologist on call at the Tampere University hospital deems the patient unable to benefit from mechanical thrombectomy

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Either verified large vessel occlusion with computed tomography angiography in Seinäjoki central hospital or positive prehospital stroke severity scale for large vessel occlusion (Finnish Prehospital Stroke Scale: FPSS) and eligibility for mechanical thrombectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference of transport times from the onset of ambulance transport to Tampere university hospital until the recording of CT Scout image | from onset of symptoms up to 24 hours
  minutes

SECONDARY OUTCOMES:
The difference of onset to revascularisation time between the groups from the onset of symptoms (last known well) until save time of "post revascularization" image | from onset of symptoms up to 24 hours
  minutes
The time difference from the onset of symptoms (last known well) until the save time of "post revascularization" image | from onset of symptoms up to 24 hours
  minutes
90 days modified Rankin scale outcome | telephone interview 90 days after mechanical thrombectomy
  mRS 0-6
Availability of the ambulance to the next emergency medical services mission in its own region. Time to next ems mission | from the beginning of ambulance transport up to 24 hours
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Sanna Hoppu, MD, PhD, Study Director — Centre of Emergency Medical Services, Tampere University Hospital
Locations (1):
- Tampere University hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided